CLINICAL TRIAL: NCT04021459
Title: Preliminary Descriptive Exploratory Pilot Study Research of Circulating Tumor Cells Released During Endometrial Cancer Surgery
Brief Title: Research of Circulating Tumor Cells Released During Endometrial Cancer Surgery.
Acronym: E-CTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RECHMPL19_0178
Record Dates: First submitted 2019-07-15; First posted 2019-07-16 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2021-09

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; circulating tumor cells; laparoscopy
MeSH Terms: conditions — Endometrial Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: women with endometrial cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- women with endometrial cancer (Other)
  Interventions: Procedure: blood samples

INTERVENTIONS:
Procedure: blood samples — 3 samples: One before surgery on the arm vein (peripheral)
  Two during the surgery, on two different venipuncture site :
  * One on the arm vein (peripheral)
  * One on ovarian vein (close to the tumor) All samples will be tested by the CellSearch method.

SUMMARY:
The purpose of this study is to investigate the spread of Circulating Tumor Cells (CTC) during surgery in endometrial cancer. Although this cancer is often discovered at early stage, the risk of recurrence is estimated at 6 to 21%, according to grade. Early stage tumor is accessible for curative surgical treatment by laparoscopy but this kind of surgery may induce CTCs spread, and could be an explanation of this recurrence. Through this study, concordance between two blood punction sites, peripheral vein and ovarian vein, will be evaluated to detect these cells during surgery.

DETAILED DESCRIPTION:
The goal of this single-center clinical trial is to determine the best blood punction site to observe the spreading of CTC during surgery in endometrial cancer. CTCs are very rare events on blood and their detection require extremely sensitive technologies. This pilot study will investigate CTC spread during surgery on 10 patients with endometrial cancer.

The main objective is to compare venipuncture site for detection of CTCs in endometrial cancer during surgery. Blood samples are collected on a simple sampling (arm) compared to sampling as close as possible to the tumor (ovarian vein).

ELIGIBILITY:
Inclusion Criteria:

* Patients with endometrial cancer
* Being affiliated or benefiting from a French social security system

Exclusion Criteria:

* Patients with an other cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment | During surgery (at the ligature of the ovarian ligament)
  Presence or not of at least one CTC during endometrial cancer surgery detected on two venipuncture site (peripheral and ovarian vein).

SECONDARY OUTCOMES:
Quantitative assessment | Before surgery and during surgery
  Number of CTC detected from each sampling

CONTACTS AND LOCATIONS:
Overall Officials: Gauthier RATHAT, PHD, Study Director — University of Montpellier
Locations (2):
- France (2):
  - Montpellier University Hospital, Montpellier
  - CHU de Nîmes, Nîmes

REFERENCES:
- [Result] Francini S, Duraes M, Rathat G, Macioce V, Mollevi C, Pages L, Ferrer C, Cayrefourcq L, Alix-Panabieres C. Circulating Tumor Cell Detection by Liquid Biopsy during Early-Stage Endometrial Cancer Surgery: A Pilot Study. Biomolecules. 2023 Feb 24;13(3):428. doi: 10.3390/biom13030428. PMID 36979364